CLINICAL TRIAL: NCT04060953
Title: Health-Related Quality of Life Measures to Optimize Chronic Pain Management
Brief Title: Quality of Life in Managing Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, John C. Licciardone, D.O., M.S., M.B.A., Principal Investigator, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300690
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health-Related Quality of Life Report (Experimental): Participants randomized to this arm will receive the Health-Related Quality of Life Report.
  Interventions: Other: Health-Related Quality of Life Report
- Wait List to Receive the Report (No Intervention): Participants randomized to this arm will receive the Health-Related Quality of Life Report following completion of the study.

INTERVENTIONS:
Other: Health-Related Quality of Life Report — Subject report and interpretation guide based on SPADE cluster scores
  Arms: Health-Related Quality of Life Report

SUMMARY:
This study evaluates the use of a health-related quality of life report based on the SPADE cluster (sleep disturbance, pain interference with activities, anxiety, depression, and low energy/fatigue) derived from the PROMIS-29 instrument in patients with chronic low back pain. Half of the participants will receive the report, while the other half will not.

DETAILED DESCRIPTION:
The health-related quality of life report provides participants with an overall score on the SPADE cluster and scores on each of its five component scales. The recently released Federal Pain Research Strategy states that pain cannot be measured in isolation, but rather should be assessed in conjunction with other outcome measures in 'non-pain domains,' such as quality of life. It recognizes that pain may be affected by, and affect, such patient attributes as sleep, mood, cognition, function, and quality of life. Further, the report states that improvement in pain without concomitant improvement in other domains may not constitute a clinically meaningful outcome. This study aims to assess the utility of a health-related quality of life report in improving quality of life, back pain intensity, and back-related disability in participants with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

Chronic Low Back Pain based on criteria established by the NIH Task Force on Research Standards for Chronic Low Back Pain AND SPADE Cluster Score ≥ 55

Exclusion Criteria:

Absence of Chronic Low Back Pain OR SPADE Cluster Score < 55

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
PROMIS-29 Quality of Life Measures | 3 Months Post-Randomization
  SPADE Cluster Score (acronym represents Sleep Disturbance, Pain Interference, Anxiety, Depression, and Low Energy/Fatigue subscales derived from the PROMIS-29). Each raw subscale score ranges from 4 to 20. Each subscale raw score is then converted to a population-normed "t-score," with a mean of 50 and standard deviation of 10. The SPADE Cluster Score is then computed as the mean of these five subscale t-scores. Higher t-scores on the SPADE Cluster and each of its component scales represent worse outcomes.

SECONDARY OUTCOMES:
Low Back Pain Intensity | 3 Months Post-Randomization
  Numerical Rating Scale for Pain (0-10).
Back-Related Disability | 3 Months Post-Randomization
  Roland-Morris Disability Questionnaire (0-24).

OTHER OUTCOMES:
Utility of the Health-Related Quality of Life Report | 1 Month Post-Randomization
  Survey of participants in the experimental treatment arm to measure the overall value of the report, various perceptions of it, and actions taken by participants in response to the report, including sharing it with their physicians or other health care providers.

CONTACTS AND LOCATIONS:
Overall Officials: John C Licciardone, DO, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No